CLINICAL TRIAL: NCT00291876
Title: Double-blind Randomized Study to Evaluate the Immunogenicity and Reactogenicity of Two Different Lots of GlaxoSmithKline Biologicals' Inactivated Hepatitis A Vaccine Containing 1440 EL.U of Antigen Per mL and Injected According to a 0, 12 Month Schedule in Healthy Adult Volunteers
Brief Title: Long-Term Immune Persistence of GlaxoSmithKline Biologicals' Inactivated Hepatitis A Vaccine Injected According to a 0, 12-month Schedule
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 100571 (M138); 100572 (M150) (Other: GSK); 100573 (M162) (Other: GSK); 100574 (M174) (Other: GSK); 100575 (M186) (Other: GSK); 110677 (M198) (Other: GSK); 110678 (M210) (Other: GSK); 110679 (Other: GSK); 110680 (Other: GSK); 110681 (Other: GSK)
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Results first posted 2010-03-08 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-01

CONDITIONS: Hepatitis A
Keywords: HAVRIX™; Hepatitis A
MeSH Terms: conditions — Hepatitis A | interventions — Hepatitis A Vaccines

ARMS (1):
- Havrix Group (Experimental): Subjects who received during the primary study 2 doses of Havrix™ at Day 0 and at Month 12.
  Interventions: Biological: Havrix™

INTERVENTIONS:
Biological: Havrix™ — 2 doses at 12 months interval

SUMMARY:
The aim of this study is to evaluate the persistence of hepatitis A antibodies at 138, 150, 162, 174,186, 198, 210, 222, 234 and 246 months after subjects received their first dose of a 2 dose vaccination schedule of hepatitis A vaccine.

This protocol posting deals with objectives & outcome measures of the extension phase at year 11 to 20.

No additional subjects will be recruited during this long-term follow-up.

DETAILED DESCRIPTION:
This is a long-term follow-up study at Years 11, 12, 13, 14, 15, 16, 17, 18, 19 and 20 after primary vaccination with GSK Biologicals' hepatitis A vaccine (two-dose schedule). To evaluate the long-term antibody persistence, volunteers will donate a blood sample at Years 11, 12, 13, 14, 15, 16, 17, 18, 19 and 20 after the first vaccine dose of the primary vaccination course to determine their anti-hepatitis A (anti-HAV) antibody concentrations.

If a subject has become seronegative for anti-HAV antibodies during any of the long-term blood sampling time point (i.e. Months 138, 150, 162, 174,186, 198, 210, 222, 234 and 246), he/ she will be offered an additional vaccine dose. A blood sample will be taken on the day of the additional vaccination 14 days and one month after additional vaccination to evaluate the immune response following this vaccination.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007 and to extend the follow up until Year 20.

The study has 10 phases: 100571, 100572, 100573, 100574, 100575, 110677, 110678, 110679, 110680, 110681.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who had received at least one dose of the study vaccine in the primary study
* Written informed consent will have been obtained from the subjects before the blood sampling visit of each year.

Ages: 29 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2004-01-01; Primary Completion 2013-03-01 (Actual); Study Completion 2013-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wilrijk, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Van Herck K, Jacquet JM, Van Damme P. Antibody persistence and immune memory in healthy adults following vaccination with a two-dose inactivated hepatitis A vaccine: long-term follow-up at 15 years. J Med Virol. 2011 Nov;83(11):1885-91. doi: 10.1002/jmv.22200. Epub 2011 Aug 23. PMID 21915861
- [Background] Van Herck K, Crasta PD, Messier M, Hardt K, Van Damme P. Seventeen-year antibody persistence in adults primed with two doses of an inactivated hepatitis A vaccine. Hum Vaccin Immunother. 2012 Mar;8(3):323-7. doi: 10.4161/hv.18617. Epub 2012 Feb 13. PMID 22327499
- [Derived] Agrawal A, Kolhapure S, Andani A, Ota MOC, Badur S, Karkada N, Mitra M. Long-Term Persistence of Antibody Response with Two Doses of Inactivated Hepatitis A Vaccine in Children. Infect Dis Ther. 2020 Dec;9(4):785-796. doi: 10.1007/s40121-020-00311-8. Epub 2020 Jul 24. PMID 32710245
- [Derived] Theeten H, Van Herck K, Van Der Meeren O, Crasta P, Van Damme P, Hens N. Long-term antibody persistence after vaccination with a 2-dose Havrix (inactivated hepatitis A vaccine): 20 years of observed data, and long-term model-based predictions. Vaccine. 2015 Oct 13;33(42):5723-5727. doi: 10.1016/j.vaccine.2015.07.008. Epub 2015 Jul 16. PMID 26190091
- [Derived] Hens N, Habteab Ghebretinsae A, Hardt K, Van Damme P, Van Herck K. Model based estimates of long-term persistence of inactivated hepatitis A vaccine-induced antibodies in adults. Vaccine. 2014 Mar 14;32(13):1507-13. doi: 10.1016/j.vaccine.2013.10.088. Epub 2014 Feb 7. PMID 24508042
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 100571 (M138) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 100571 are summarised with studies 100572, 100573, 100574, 100575, 110677, 110678, 110679, 110680, and 110681 on the GSK Clinical Study
- Available data/document: Informed Consent Form: 100571 (M138) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 100571 (M138) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 100571 (M138) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 100571 (M138) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 100571 (M138) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant Flow and Baseline Measures are given for each of the follow-up time points- Months 138, 150, 162, 174, 186, 198, 210, 222, 234 and 246. Note that not all subjects returned and participated in each of the intermediate follow-up time points.
Pre-assignment Details: The Long-Term (LT) Total Cohort included all subjects who returned for the follow-up and who belonged to the Total Cohort in the primary study.
  The Long Term According-to-Protocol (LT-ATP) cohort for immunogenicity included subjects who returned for the follow-up and who were included in the ATP cohort for immunogenicity of the primary study.
Period: Month 138
Arm/Group | Havrix Group
Started | 107
Completed | 107
Not Completed | 0
Period: Month 150
Arm/Group | Havrix Group
Started | 117
Completed | 117
Not Completed | 0
Period: Month 162
Arm/Group | Havrix Group
Started | 127
Completed | 127
Not Completed | 0
Period: Month 174
Arm/Group | Havrix Group
Started | 127
Completed | 127
Not Completed | 0
Period: Month 186
Arm/Group | Havrix Group
Started | 129
Completed | 129
Not Completed | 0
Period: Month 198
Arm/Group | Havrix Group
Started | 135
Completed | 135
Not Completed | 0
Period: Month 210
Arm/Group | Havrix Group
Started | 124
Completed | 124
Not Completed | 0
Period: Month 222
Arm/Group | Havrix Group
Started | 114
Completed | 114
Not Completed | 0
Period: Month 234
Arm/Group | Havrix Group
Started | 110
Completed | 110
Not Completed | 0
Period: Month 246
Arm/Group | Havrix Group
Started | 116
Completed | 116
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline Measures are given for each of the follow-up time points- Months 138, 150, 162, 174, 186, 198, 210, 222, 234 and 246. Note that not all subjects returned and participated in each of the intermediate follow-up time points.
Arm/Group | Havrix Group
Number analyzed (Participants) | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Month 138 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Years
    number analyzed (Participants) | 107
    (all) | 42.2 (5.44)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Month 150 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Years
    number analyzed (Participants) | 117
    (all) | 42.9 (5.35)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Month 162 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Years
    number analyzed (Participants) | 127
    (all) | 43.4 (5.34)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Month 174 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Years
    number analyzed (Participants) | 127
    (all) | 44.5 (5.37)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Month 186 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Years
    number analyzed (Participants) | 129
    (all) | 45.4 (5.39)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Month 198 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Years | 46.3 (5.35)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Month 210 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Years
    number analyzed (Participants) | 124
    (all) | 47.6 (5.39)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Month 222 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Years
    number analyzed (Participants) | 114
    (all) | 48.5 (5.39)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Month 234 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Years
    number analyzed (Participants) | 110
    (all) | 49.6 (5.42)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Month 246 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Years
    number analyzed (Participants) | 116
    (all) | 50.8 (5.34)
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Month 138 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Participants
    number analyzed (Participants) | 107
    Female | 77
    Male | 30
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Month 150 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Participants
    number analyzed (Participants) | 117
    Female | 87
    Male | 30
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Month 162 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Participants
    number analyzed (Participants) | 127
    Female | 93
    Male | 34
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Month 174 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Participants
    number analyzed (Participants) | 127
    Female | 94
    Male | 33
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Month 186 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Participants
    number analyzed (Participants) | 129
    Female | 98
    Male | 31
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Month 198 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Participants
    Female | 103
    Male | 32
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Month 210 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Participants
    number analyzed (Participants) | 124
    Female | 93
    Male | 31
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Month 222 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Participants
    number analyzed (Participants) | 114
    Female | 83
    Male | 31
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Month 234 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Participants
    number analyzed (Participants) | 110
    Female | 81
    Male | 29
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Month 246 Population: Note that not all subjects returned and participated in each of the intermediate follow-up time points.
  Participants
    number analyzed (Participants) | 116
    Female | 86
    Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Anti-hepatitis A Virus (Anti-HAV) Antibody Concentration
Description: Concentrations given as geometric mean concentration (GMC) expressed as milli-international unit per millilitre (mIU/mL). ** = Regarding Month 234 data, please note that there were 5 subjects for whom serum sample tube was broken and thus due to risk of contamination the test were not performed. Hence these subjects were not included in the LT-ATP cohort for immunogenicity analysis at Month 234. $ = Regarding Month 246 data, please note there was 1 subject for whom serum sample tube was broken and hence scrapped by laboratory. Hence this subject was not included in the LT-ATP cohort for immunogenicity analysis at Month 246.
Time Frame: At Months 138, 150, 162, 174, 186, 198, 210, 222, 234 and 246
Population: Analysis was performed on the Long Term According-to-Protocol (LT-ATP) cohort for analysis of immunogenicity, on subjects with available data for the defined timepoint.
  * The laboratory assay was changed at Month 138, thus the blood samples were re-tested with the old assay for the sake of bridging.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Havrix Group
Number analyzed (Participants) | 102
mIU/mL
  Month 138 (N=79) | 748.1 [614.3 to 911.1]
  Month 138 (N=85)* | 378.6 [304.3 to 471.0]
  Month 150 (N=93) | 419.3 [335.1 to 524.8]
  Month 162 (N=101) | 342.2 [270.8 to 432.5]
  Month 174 (N=102) | 318.9 [257.0 to 395.5]
  Month 186 (N=98) | 353.1 [284.0 to 439.1]
  Month 198 (N=101) | 339.9 [273.2 to 422.9]
  Month 210 (N=91) | 369.3 [294.0 to 463.9]
  Month 222 (N=86) | 340.1 [271.1 to 426.7]
  Month 234 (N=79)** | 283.3 [222.4 to 361.0]
  Month 246 (N=85)$ | 317.3 [247.4 to 407.1]

2. Primary Outcome: Number of Seropositive Subjects Against Hepatitis A Virus
Description: A seropositive subject was a vaccinated subject whose concentrations for antibodies against hepatitis A virus (anti-HAV) were equal or above (>=) the assay cut-off for seropositivity of 15 milli-international units per milliliter (mIU/mL). ** = Regarding Month 234 data, please note that there were 5 subjects for whom serum sample tube was broken and thus due to risk of contamination the test were not performed. Hence these subjects were not included in the LT-ATP cohort for immunogenicity analysis at Month 234. $ = Regarding Month 246 data, please note there was 1 subject for whom serum sample tube was broken and hence scrapped by laboratory. Hence this subject was not included in the LT-ATP cohort for immunogenicity analysis at Month 246.
Time Frame: At Months 138, 150, 162, 174, 186, 198, 210, 222, 234 and 246
Population: Analysis was performed on the Long Term According-to-Protocol (LT-ATP) cohort for analysis of immunogenicity, on subjects with available data for the defined timepoint. *The laboratory assay was changed at Month 138, thus the blood samples were re-tested with the old assay for the sake of bridging.
Measure: Number; unit: Subjects
Arm/Group | Havrix Group
Number analyzed (Participants) | 102
Subjects
  Month 138 (N=79) | 77
  Month 138 (N=85)* | 82
  Month 150 (N=93) | 90
  Month 162 (N=101) | 98
  Month 174 (N=102) | 100
  Month 186 (N=98) | 95
  Month 198 (N=101) | 97
  Month 210 (N=91) | 88
  Month 222 (N=86) | 86
  Month 234 (N=79)** | 79
  Month 246 (N=85)$ | 85

3. Secondary Outcome: Anti-hepatitis A Virus (Anti-HAV) Antibody Concentration
Description: Concentrations given as GMC expressed as mIU/mL. 4 subjects received additional vaccination at Month 186 and 1 subject at Month 198.
  Please note that value 14.9 means <15.
Time Frame: Before additional vaccination, 14 days after additional vaccination and 30 days after additional vaccination
Population: Analysis was performed on the Long Term Total cohort, only on subjects who received an additional vaccine dose during the current long-term follow-up study. If a subject became seronegative (< 15 mIU/mL) at any of the long-term blood sampling timepoint, he/she was offered an additional vaccine dose.
Measure: Number; unit: mIU/mL
Arm/Group | Havrix Group
Number analyzed (Participants) | 5
mIU/mL
  Subject 1 Month 186 before | 14.9
  Subject 1 Month 186 day 14 | 15
  Subject 1 Month 186 day 30 | 26
  Subject 2 Month 186 before | 14.9
  Subject 2 Month 186 day 14 | 453
  Subject 2 Month 186 day 30 | 787
  Subject 3 Month 186 before | 15
  Subject 3 Month 186 day 14 | 3102
  Subject 3 Month 186 day 30 | 3819
  Subject 4 Month 186 before | 16
  Subject 4 Month 186 day 14 | 1636
  Subject 4 Month 186 day 30 | 2051
  Subject 5 Month 198 before | 16
  Subject 5 Month 198 day 14 | 3222
  Subject 5 Month 198 day 30 | 4894

4. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. Additional vaccination was given to 4 subjects at the Month 186 timepoint and to 1 subject at the Month 198 timepoint.
Time Frame: During the 4-day (Days 0-3) follow-up period after additional vaccination
Population: as for outcome 3
Measure: Number; unit: subjects
Arm/Group | Havrix Group
Number analyzed (Participants) | 5
subjects
  Pain Month 186 (N=4) | 2
  Redness Month 186 (N=4) | 0
  Swelling Month 186 (N=4) | 0
  Pain Month 198 (N=1) | 1
  Redness Month 198 (N=1) | 0
  Swelling Month 198 (N=1) | 0

5. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include fatigue, fever, gastrointestinal symptoms and headache.
  4 subjects received additional vaccination at Month 186 and 1 subject at Month 198.
Time Frame: During the 4-day (Days 0-3) follow-up period after additional vaccination
Population: as for outcome 3
Measure: Number; unit: subjects
Arm/Group | Havrix Group
Number analyzed (Participants) | 5
subjects
  Fatigue Month 186 (N=4) | 2
  Fever Month 186 (N=4) | 0
  Gastrointestinal Month 186 (N=4) | 1
  Headache Month 186 (N=4) | 1
  Fatigue Month 198 (N=1) | 0
  Fever Month 198 (N=1) | 0
  Gastrointestinal Month 198 (N=1) | 0
  Headache Month 198 (N=1) | 0

6. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  4 subjects received additional vaccination at Month 186 and 1 at Month 198.
Time Frame: During the 30-day follow-up period after additional vaccination
Population: as for outcome 3
Measure: Number; unit: subjects
Arm/Group | Havrix Group
Number analyzed (Participants) | 5
subjects
  Month 186 (N=4) | 0
  Month 198 (N=1) | 0

7. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE) Assessed by the Investigator as Related to Primary Study Vaccination, Procedures or Lack of Vaccine Efficacy
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above
Time Frame: At Months 138, 150, 162, 174, 186, 198, 210, 222, 234 and 246
Population: Analysis was performed on the Long Term Total cohort, on subjects with available data for the defined timepoint.
Measure: Number; unit: Subjects
Arm/Group | Havrix Group
Number analyzed (Participants) | 135
Subjects
  Month 138 (N=107) | 0
  Month 150 (N=117) | 0
  Month 162 (N=127) | 0
  Month 174 (N=127) | 0
  Month 186 (N=129) | 0
  Month 198 (N=135) | 0
  Month 210 (N=124) | 0
  Month 222 (N=114) | 0
  Month 234 (N=110) | 0
  Month 246 (N=116) | 0

8. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE) After Additional Vaccination
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
  4 subjects received additional vaccination at Month 186 and 1 at Month 198.
Time Frame: During the 30-day follow-up period after additional vaccination
Population: as for outcome 3
Measure: Number; unit: subjects
Arm/Group | Havrix Group
Number analyzed (Participants) | 5
subjects
  Month 186 (N=4) | 0
  Month 198 (N=1) | 0

9. Secondary Outcome: Number of Subjects Reporting Pregnancies After Additional Vaccination
Description: The number of subjects with outcome of pregnancies reported among subjects who had received the additional vaccination was tabulated. 4 subjects received additional vaccination at Month 186 and 1 subject at Month 198.
Time Frame: At Months 186 and 198
Population: as for outcome 3
Measure: Number; unit: Subject
Arm/Group | Havrix Group
Number analyzed (Participants) | 5
Subject
  Subjects with pregnancy - At Month 186 (N=4) | 0
  Subjects with pregnancy - At Month 198 (N=1) | 0

ADVERSE EVENTS:
Time Frame: SAEs: At Months 138, 150, 162, 174, 186, 198, 210, 222 234 and 246. Other adverse events: within the 4-day periods after additional vaccination (at Month 186 or 198), only in subjects who received additional vaccination at the specified time point.
Description: Analyses were performed on the Long-Term (LT) Total Cohort which included all subjects who returned for the follow-up and who belonged to the Total Cohort in the primary study. Maximum amount of subjects which participated at Month 198 has been taken as the number of subjects at risk for SAEs.
Arm/Group | Havrix Group
Serious Adverse Events (participants affected / at risk) | 0/135
Other Adverse Events (participants affected / at risk) | 2/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Havrix Group (N=5)
Pain (General disorders) | 2/4 — Occurrence of the specified adverse event collected 4-days after additional dose reported among the 4 subjects receiving vaccination at Month 186
Pain (General disorders) | 1/1 — Occurrence of the specified adverse event collected 4-days after additional dose reported by the 1 subject receiving vaccination at Month 198
Fatigue (General disorders) | 2/4 — Occurrence of the specified adverse event collected 4-days after additional dose reported among the 4 subjects receiving vaccination at Month 186
Gastrointestinal (General disorders) | 1/4 — Occurrence of the specified adverse event collected 4-days after additional dose reported among the 4 subjects receiving vaccination at Month 186
Headache (General disorders) | 1/4 — Occurrence of the specified adverse event collected 4-days after additional dose reported among the 4 subjects receiving vaccination at Month 186

LIMITATIONS AND CAVEATS:
For 5 subjects at Month 234, serum sample tubes were broken. Due to risk of contamination, anti-HAV concentrations analyses were not performed for these subjects, who were excluded in the LT-ATP cohort for immunogenicity analysis at Month 234.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.